CLINICAL TRIAL: NCT04858802
Title: The EXPAND Study: A Clinical Evaluation of PROPEL® Contour Sinus Implant Placement in the Frontal Sinus Ostium Following In-office Bilateral Balloon Dilation
Brief Title: A Clinical Evaluation of PROPEL® Contour Sinus Implant
Acronym: EXPAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P500-1220
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Frontal Sinus; Balloon Dilation
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Intrapatient control in which eligible subjects will receive the PROPEL Contour Sinus Implant (Treatment) on one side, and no implant (Control) on the contralateral side.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PROPEL Contour Sinus Implant (Experimental): Following successful in-office bilateral balloon dilation, placement of PROPEL Contour Sinus Implant in the randomized side.
  Interventions: Device: PROPEL Contour Sinus Implant
- Balloon Sinus Dilation Alone (Active Comparator): Following successful in-office bilateral balloon dilation, placement of no implant on the contralateral side.
  Interventions: Procedure: Balloon Sinus Dilation Alone

INTERVENTIONS:
Device: PROPEL Contour Sinus Implant — 370 mcg mometasone furoate-coated sinus implant
  Arms: PROPEL Contour Sinus Implant
Procedure: Balloon Sinus Dilation Alone — No PROPEL Contour Sinus Implant
  Arms: Balloon Sinus Dilation Alone

SUMMARY:
The objective of this study is to evaluate the efficacy of PROPEL Contour placement following an in-office frontal sinus balloon dilation (SBD) in patients with chronic rhinosinusitis (CRS)

DETAILED DESCRIPTION:
A post-market, randomized, intra-patient controlled, blinded multicenter study with 80 randomized subjects at up to 20 study centers.

After successful in-office bilateral balloon dilation of the frontal sinus ostium (FSO) using the VenSure™ Nav Balloon Device and Fiagon Cube Navigation System, patients will be randomized to receive one PROPEL Contour Sinus Implant on one side while the contralateral side serves as the control.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older.
2. Patient is willing and able to comply with protocol requirements.
3. Patient has confirmed diagnosis of CRS per International Consensus Statement on Allergy and Rhinology, Rhinosinusitis 2021 (ICAR:RS) guidelines.
4. Bilateral disease in the frontal sinuses (Lund-Mackay CT score of ≥1 on each side) on CT scan within 90 days prior to the baseline.
5. A successfully completed in-office bilateral balloon dilation of the FSO with no complication on either side that, in the opinion of the clinical investigator is amenable for PROPEL Contour Sinus Implant placement in both FSO

Exclusion Criteria:

1. Patient has structural obstruction that precludes endoscopic visualization of one or both FSOs prior to implant placement.
2. Expanded amount of ethmoid sinonasal polyps extending beyond the middle meatus (grade > 2) unless reduced 30 days prior to the baseline procedure
3. Oral-steroid dependent condition such as chronic obstructive pulmonary disease (COPD) or other conditions.
4. Known history of allergy or intolerance to corticosteroids or mometasone furoate.
5. Patients with a known hypersensitivity to lactide, glycolide or caprolactone copolymers.
6. Patients with electronic devices in direct connection to the brain or the nervous system such as implantable neurostimulators (e.g. deep brain stimulation), programmable cerebrospinal fluid (CSF) shunts.
7. Patients with monopolar pacemakers (older designs, with lower resistance to interference) or ICD's (implantable cardioverter defibrillator).
8. Patients with implantable, body worn devices such as insulin pumps.
9. Evidence of purulence coming from paranasal sinuses or ostiomeatal complex.
10. Clinical evidence of acute bacterial sinusitis or invasive fungal sinusitis (e.g. bone erosion on prior CT scan, necrotic sinus tissue).
11. Active viral illness (e.g., flu, shingles).
12. Use of parenteral or injected steroids (e.g. Kenalog) 30 days prior to the baseline procedure.
13. Use of oral steroids, budesonide or other sinus steroid irrigations/rinses or drops, nebulized steroids administered nasally 14 days prior to baseline procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Sacramento ENT/DaVinci Research, LLC, Sacramento, California
  - San Francisco Otolaryngology, San Francisco, California
  - ENT & Allergy Associate of Florida, LLC, Boca Raton, Florida
  - ENT & Allergy Associate of Florida, LLC, Boynton Beach, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Ascentist Physicians Group, Leawood, Kansas
  - Kentuckiana Ear, Nose & Throat PSC, Louisville, Kentucky
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Madison ENT, New York, New York
  - Ohio Sinus Institute, Dublin, Ohio
  - Fort Worth ENT & Sinus, Fort Worth, Texas
  - Collin County ENT, Frisco, Texas
  - ENT Associates of Texas, McKinney, Texas
  - Alamo ENT Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from fourteen locations in the United States.
Pre-assignment Details: A total of 89 patients were assessed for eligibility. Eight patients did not meet inclusion criteria or met exclusion criteria. One patient withdrew from the study prior to randomization. A total of 80 patients met final eligibility and were randomized.
Units Other Than Participants: sinus sides
Period: Overall Study
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Started | 80; 80 sinus sides | 80; 80 sinus sides
Completed Day 45 Follow-up Visit | 80; 80 sinus sides | 80; 80 sinus sides
Completed | 78; 78 sinus sides | 78; 78 sinus sides
Not Completed | 2; 2 sinus sides | 2; 2 sinus sides
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Following successful in-office bilateral balloon dilation, placement of PROPEL Contour Sinus Implant in the frontal sinus ostium occurred on the randomized side. The opposing side served as control.
  PROPEL Contour Sinus Implant: 370 mcg mometasone furoate-coated sinus implant
Arm/Group | All Participants
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.38)
Sex/Gender, Customized [Number; unit: participants]
  Female | 30
  Male | 50
Race/Ethnicity, Customized [Number; unit: participants]
  White | 69
  Asian | 7
  Black or African American | 2
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 80
Number of prior endoscopic sinus surgeries (ESS) [Number; unit: participants]
  0 | 36
  1 | 26
  2 | 12
  3 | 4
  ≥ 4 | 2
Asthma diagnosed by physician [Number; unit: participants] — Asthma severity was assessed as either mild, moderate, or severe by clinical investigator.
  participants
    Yes, any severity | 15
    Yes, mild | 13
    Yes, moderate | 2
    Yes, severe | 0
Allergic rhinitis diagnosed by physician [Number; unit: participants] — Allergic rhinitis severity was assessed as either mild, moderate, or severe by clinical investigator.
  participants
    Yes, any severity | 68
    Yes, mild | 39
    Yes, moderate | 27
    Yes, severe | 2
Aspirin intolerance or allergy [Number; unit: participants] | 2
Lund-Mackay score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay scale is used as a staging system for chronic rhinosinusitis. A score is assigned by the grader based on the opacification of anatomical regions of the paranasal sinuses as visualized on CT imaging. The grader assigns a value of 0 if the region is totally patent, 1 if it is partially opacified, or 2 if it is completely opacified. The regions evaluated are the frontal, anterior ethmoid, posterior ethmoid, maxillary, and sphenoid sinuses. The ostiomeatal complex (OMC) is scored either 0 or 2. The maximum score for each side is thus 12, with a total score determined out of 24.
  units on a scale
    Total score (left + right) | 9.21 (3.83)
    Frontal sinus score (left + right) | 2.19 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: Difference in FSO Patency by Blinded Reviewer
Description: Side-to-side difference in frontal sinus ostium (FSO) patency at Day 45 based on cross-sectional area of FSO by computed tomography (CT) measurements performed by an independent, blinded reviewer. Cross-sectional area of FSO was measured via computer-assisted segmentation of CT images.
Time Frame: Day 45
Population: Number of units (sinus sides) analyzed represents number of participants with data evaluable.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 76 | 76
mm^2 | 16.54 (20.83) | 12.36 (16.10)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; The null hypothesis was that there would no difference in FSO cross-sectional area between treatment and control sides at Day 45; Test type: Superiority; p = 0.059, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Net) = 4.19, 95% CI 2-sided [-0.2 to 8.6], Standard Deviation 19.08 — Difference = PROPEL Contour Sinus Implant mean FSO cross-sectional area minus balloon sinus dilation alone mean FSO cross-sectional area

2. Secondary Outcome: FSO Cross-sectional Area Change From Baseline on CT by an Independent, Blinded Reviewer
Description: FSO cross-sectional area change from baseline to Day 45 and change from baseline to Day 180 per CT assessment performed by an independent, blinded reviewer. FSO cross-sectional area was measured via computer-assisted segmentation of CT images.
Time Frame: Baseline, Day 45, and Day 180
Population: Number of units (sinus sides) analyzed represents number of participants with data evaluable for the corresponding timepoint.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 75 | 75
mm^2
  Change from baseline to Day 45 | 2.63 (9.95) | 1.15 (11.09)
  Change from baseline to Day 180 | 3.20 (10.97) | 5.95 (13.78)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.328, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-1.5 to 4.5], Standard Deviation 12.98 — Difference = PROPEL Contour Sinus Implant mean FSO cross-sectional area change from baseline to Day 45 minus balloon sinus dilation alone mean FSO cross-sectional area change from baseline to Day 45
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.063, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -2.75, 95% CI 2-sided [-5.7 to 0.2], Standard Deviation 12.64 — Difference = PROPEL Contour Sinus Implant mean FSO cross-sectional area change from baseline to Day 180 minus balloon sinus dilation alone mean FSO cross-sectional area change from baseline to Day 180

3. Secondary Outcome: CT Frontal Sinus Outflow Tract (FSOT) Volume by Blinded Reviewer
Description: FSOT, referring to the region of the frontal sinus surrounding the FSO, bordered superiorly by the frontal infundibulum and inferiorly by the frontal recess, is assessed by blinded reviewer. FSOT volume was measured via computer-assisted segmentation of CT images.
Time Frame: Days 45 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 76 | 76
mm^3
  Day 45 | 383.11 (437.19) | 332.17 (399.68)
  Day 180: number analyzed (sinus sides) | 75 | 75
  Day 180 | 386.86 (413.56) | 414.30 (427.56)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.306, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 50.94, 95% CI 2-sided [-47.5 to 149.4], Standard Deviation 430.80 — Difference = PROPEL Contour Sinus Implant mean FSOT volume minus balloon sinus dilation alone mean FSOT volume
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.567, t-test, 2 sided; Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -27.44, 95% CI 2-sided [-122.5 to 67.6], Standard Deviation 413.22 — Difference = PROPEL Contour Sinus Implant mean FSOT volume minus balloon sinus dilation alone mean FSOT volume

4. Secondary Outcome: CT FSO Minimum Diameter by Blinded Reviewer
Description: CT FSO minimum diameter assessed by blinded independent reviewer to assess extent of the disease in the frontal sinuses. FSO minimum diameter was measured via computer-assisted segmentation of CT images.
Time Frame: Days 45 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 76 | 76
mm
  Day 45 | 2.38 (1.94) | 1.89 (1.79)
  Day 180: number analyzed (sinus sides) | 75 | 75
  Day 180 | 2.56 (2.23) | 2.54 (2.13)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.031, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Net) = 0.48, 95% CI 2-sided [0.0 to 0.9], Standard Deviation 1.92 — Difference = PROPEL Contour Sinus Implant mean FSO minimum diameter minus balloon sinus dilation alone mean FSO minimum diameter
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.943, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.5 to 0.5], Standard Deviation 2.27 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: CT Zinreich's Modified Lund-Mackay Score for the Frontal Sinus by Blinded Reviewer
Description: CT Zinreich's modified Lund-Mackay score for the frontal sinus assessed by blinded independent reviewer to assess extent of the disease in the frontal sinuses.
  Zinreich's modified Lund-Mackay scale ranges from 0 to 5. Higher scores indicate a worse outcome.
Time Frame: Days 45 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 78 | 78
score on a scale
  Day 45 | 1.23 (1.22) | 1.28 (1.38)
  Day 180 | 1.22 (1.40) | 1.05 (1.27)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.715, t-test, 2 sided; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.3 to 0.2], Standard Deviation 1.24 — Difference = PROPEL Contour Sinus Implant mean Zinreich's modified Lund-Mackay score for the frontal sinus minus balloon sinus dilation alone mean Zinreich's modified Lund-Mackay score for the frontal sinus
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.129, t-test, 2 sided; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.0 to 0.4], Standard Deviation 0.96 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Number of Sinus Sides Requiring Post-operative Intervention by Clinical Investigators
Description: Need for post-operative intervention as determined by clinical investigators per endoscopy.
Time Frame: Days 21, 45, 90 and 180
Population: as for outcome 2
Measure: Count of Units; unit: sinus sides
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 80 | 80
sinus sides
  Day 21 | 5 | 5
  Day 45 | 14 | 17
  Day 90 | 12 | 16
  Day 180 | 12 | 16
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 1.00, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.28 to 3.60]
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.453, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.36 to 1.73]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 0.219, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.31 to 1.61]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.289, t-test, 2 sided; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.31 to 1.61]

7. Secondary Outcome: CT Cross-sectional Area of FSO by Blinded Reviewer
Description: CT cross-sectional area of FSO assessed by blinded independent reviewer to assess extent of the disease in the frontal sinuses. Cross-sectional area of FSO was measured via computer-assisted segmentation of CT images.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 75 | 75
mm^2 | 17.72 (21.05) | 17.81 (19.96)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.971, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-4.9 to 4.8], Standard Deviation 21.12 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: CT Lund-Mackay Score for the Frontal Sinus by Blinded Reviewer
Description: CT Lund-Mackay score for the frontal sinus assessed by blinded independent reviewer to assess extent of the disease in the frontal sinuses.
  The Lund-Mackay scale ranges from 0 to 2. Higher scores indicate a worse outcome.
Time Frame: Days 45 and 180
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 78 | 78
score on a scale
  Day 45 | 0.77 (0.48) | 0.77 (0.56)
  Day 180 | 0.72 (0.56) | 0.67 (0.55)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 1.00, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.1 to 0.1], Standard Deviation 0.56; Difference = PROPEL Contour Sinus Implant mean Lund-Mackay score for the frontal sinus at Day 45 minus balloon sinus dilation alone mean Lund-Mackay score for the frontal sinus at Day 45
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.288, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.0 to 0.1], Standard Deviation 0.42 — Difference = PROPEL Contour Sinus Implant mean Lund-Mackay score for the frontal sinus at Day 180 minus balloon sinus dilation alone mean Lund-Mackay score for the frontal sinus at Day 180

9. Secondary Outcome: CT Lund-Mackay Score for the Frontal Sinus by Clinical Investigators
Description: CT Lund-Mackay for the frontal sinus assessed by blinded independent reviewer to assess extent of the disease in the frontal sinuses.
  The Lund-Mackay scale ranges from 0 to 2. Higher scores indicate a worse outcome.
Time Frame: Days 45 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 79 | 79
score on a scale
  Day 45 | 0.59 (0.59) | 0.68 (0.59)
  Day 180: number analyzed (sinus sides) | 78 | 78
  Day 180 | 0.53 (0.64) | 0.59 (0.63)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.225, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.2 to 0.1], Standard Deviation 0.64 — Difference = PROPEL Contour Sinus Implant mean Lund-Mackay score for the frontal sinus at Day 45 minus balloon sinus dilation alone mean Lund-Mackay score for the frontal sinus at Day 45
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.388, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.2 to 0.1], Standard Deviation 0.65 — Difference = PROPEL Contour Sinus Implant mean Lund-Mackay score for the frontal sinus at Day 180 minus balloon sinus dilation alone modified Lund-Mackay score for the frontal sinus at Day 180

10. Secondary Outcome: Adhesion/Scarring Grade in the Frontal Recess/FSO by Clinical Investigators
Description: Endoscopic grading of adhesion/scarring grade in the frontal recess/FSO by clinical investigators.
  The adhesion/scarring grade in the frontal recess/FSO scale ranges from 0 to 4. Higher scores indicate a worse outcome.
Time Frame: Days 21, 45, 90 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 76 | 75
score on a scale
  Day 21: number analyzed (sinus sides) | 52 | 51
  Day 21 | 0.37 (0.63) | 0.41 (0.61)
  Day 45: number analyzed (sinus sides) | 60 | 60
  Day 45 | 0.30 (0.62) | 0.48 (0.75)
  Day 90: number analyzed (sinus sides) | 70 | 69
  Day 90 | 0.21 (0.54) | 0.48 (0.78)
  Day 180 | 0.24 (0.56) | 0.45 (0.74)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 0.537, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.2 to 0.1], Standard Deviation 0.68 — Difference = PROPEL Contour Sinus Implant mean adhesion/scarring grade in the frontal recess/FSO minus balloon sinus dilation alone mean adhesion/scarring grade in the frontal recess/FSO
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.010, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.3 to 0.0], Standard Deviation 0.54 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 0.003, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.4 to -0.1], Standard Deviation 0.70 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.007, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.4 to -0.1], Standard Deviation 0.66 — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Inflammation Score in the Frontal Recess/FSO by Clinical Investigators
Description: Endoscopic grading of inflammation score in the frontal recess/FSO by clinical investigators.
  Inflammation score in the frontal recess/FSO ranges from 0 to 100. Higher scores indicate a worse outcome.
Time Frame: Days 21, 45, 90 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 76 | 74
score on a scale
  Day 21: number analyzed (sinus sides) | 50 | 48
  Day 21 | 25.94 (29.31) | 28.85 (30.86)
  Day 45: number analyzed (sinus sides) | 60 | 60
  Day 45 | 19.17 (27.68) | 26.67 (32.16)
  Day 90: number analyzed (sinus sides) | 70 | 69
  Day 90 | 21.97 (34.10) | 28.62 (33.80)
  Day 180 | 17.30 (31.45) | 24.46 (33.45)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 0.634, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-12.8 to 7.9], Standard Deviation 35.55 — Difference = PROPEL Contour Sinus Implant mean inflammation score in the frontal recess/FSO minus balloon sinus dilation alone mean inflammation score in the frontal recess/FSO
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.048, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -7.63, 95% CI 2-sided [-15.2 to -0.1], Standard Deviation 29.04 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 0.028, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -7.78, 95% CI 2-sided [-14.7 to -0.9], Standard Deviation 28.79 — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.041, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -6.76, 95% CI 2-sided [-13.2 to -0.3], Standard Deviation 27.99 — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Polypoid Edema in the Frontal Recess/FSO by Clinical Investigators
Description: Endoscopic grading of polypoid edema in the frontal recess/FSO by clinical investigators.
  Polypoid edema in the frontal recess/FSO scale ranges from 0 to 3. Higher scores indicate a worse outcome.
Time Frame: Days 21, 45, 90 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 77 | 75
score on a scale
  Day 21: number analyzed (sinus sides) | 51 | 50
  Day 21 | 0.63 (0.82) | 0.88 (1.04)
  Day 45: number analyzed (sinus sides) | 60 | 61
  Day 45 | 0.53 (0.87) | 0.77 (1.01)
  Day 90: number analyzed (sinus sides) | 70 | 69
  Day 90 | 0.53 (0.93) | 0.80 (1.02)
  Day 180 | 0.52 (0.85) | 0.71 (0.93)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 0.063, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.5 to 0.0], Standard Deviation 0.96 — Difference = PROPEL Contour Sinus Implant mean polypoid edema grade in the frontal recess/FSO minus balloon sinus dilation alone mean polypoid edema grade in the frontal recess/FSO
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.015, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.4 to -0.1], Standard Deviation 0.77 — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 0.007, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.4 to -0.1], Standard Deviation 0.78 — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.034, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.4 to 0.0], Standard Deviation 0.75 — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Adhesion/Scarring Grade in the Ethmoid Sinus by Clinical Investigators
Description: Endoscopic grading of adhesion/scarring grade in the ethmoid sinus by clinical investigators.
  The adhesion/scarring grade in the ethmoid sinus scale ranges from 0 to 4. Higher scores indicate a worse outcome.
Time Frame: Day 21, 45, 90, and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 77 | 75
score on a scale
  Day 21: number analyzed (sinus sides) | 50 | 50
  Day 21 | 0.28 (0.67) | 0.30 (0.71)
  Day 45: number analyzed (sinus sides) | 62 | 62
  Day 45 | 0.34 (0.72) | 0.35 (0.73)
  Day 90: number analyzed (sinus sides) | 68 | 67
  Day 90 | 0.26 (0.66) | 0.39 (0.74)
  Day 180 | 0.29 (0.78) | 0.39 (0.75)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 0.830, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.2 to 0.2], Standard Deviation 0.65 — Difference = PROPEL Contour Sinus Implant mean adhesion/scarring grade in the ethmoid sinus minus balloon sinus dilation alone mean adhesion/scarring grade in the ethmoid sinus
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.829, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.2 to 0.1], Standard Deviation 0.59 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 0.132, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.3 to 0.0], Standard Deviation 0.64 — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.310, t-test, 2 sided; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.3 to 0.1], Standard Deviation 0.79 — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Polyp Grade in the Ethmoid Sinus by Clinical Investigators
Description: Endoscopic grading of polyp grade in the ethmoid sinus by clinical investigators.
  Polyp grade in the ethmoid sinus scale ranges from 0 to 3. Higher scores indicate a worse outcome.
Time Frame: Days 21, 45, 90 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 80 | 80
Number analyzed (sinus sides) | 77 | 77
score on a scale
  Day 21: number analyzed (sinus sides) | 51 | 51
  Day 21 | 0.29 (0.65) | 0.32 (0.62)
  Day 45: number analyzed (sinus sides) | 62 | 62
  Day 45 | 0.30 (0.61) | 0.34 (0.66)
  Day 90: number analyzed (sinus sides) | 70 | 70
  Day 90 | 0.31 (0.72) | 0.39 (0.73)
  Day 180 | 0.29 (0.64) | 0.31 (0.64)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 0.666, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.2 to 0.1], Standard Deviation 0.48 — Difference = PROPEL Contour Sinus Implant mean polyp grade in the ethmoid sinus minus balloon sinus dilation alone mean polyp grade in the ethmoid sinus
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.497, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.2 to 0.1], Standard Deviation 0.46 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 0.235, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.2 to 0.0], Standard Deviation 0.50 — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.677, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.1 to 0.1], Standard Deviation 0.41 — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: CRS Side-specific Symptom Score by Subject
Description: Subject-reported outcome of chronic rhinosinusitis (CRS) side-specific symptom score.
  The chronic rhinosinusitis side-specific symptom score scale ranges from 0 to 30. Higher scores indicate a worse outcome.
Time Frame: Days 21, 45, 90 and 180
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 79 | 79
Number analyzed (sinus sides) | 77 | 76
score on a scale
  Day 21: number analyzed (sinus sides) | 52 | 52
  Day 21 | 6.19 (4.74) | 6.25 (4.95)
  Day 45: number analyzed (sinus sides) | 60 | 60
  Day 45 | 4.75 (3.77) | 4.68 (3.90)
  Day 90: number analyzed (sinus sides) | 69 | 69
  Day 90 | 4.42 (4.21) | 4.42 (4.46)
  Day 180 | 3.86 (4.32) | 4.22 (4.76)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 21; Test type: Superiority; p = 0.868, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.7 to 0.6], Standard Deviation 2.48 — Difference = PROPEL Contour Sinus Implant mean CRS side-specific symptom total score minus balloon sinus dilation alone mean CRS side-specific symptom total score
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.823, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.5 to 0.7], Standard Deviation 2.30 — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 90; Test type: Superiority; p = 1.00, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.5 to 0.5], Standard Deviation 2.26 — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.188, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.8 to 0.2], Standard Deviation 2.16 — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: SNOT-22 Score by Subject
Description: Subject-reported outcome of SNOT-22 score.
  The Sino-Nasal Outcome Test, 22 item (SNOT-22) is a validated, disease-specific, symptom-scoring instrument consisting of 22 questions, each scored by the patient on a 6-point scale, ranging from a score of 0 ("no problem") to 5 ("problem as bad as it can be"). The maximum total score for all symptoms is equal to 110.
  Higher scores indicate a worse outcome.
Time Frame: Day 180
Population: Number of units (sinus sides) analyzed represents number of participants with data evaluable.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 79 | 79
Number analyzed (sinus sides) | 77 | 77
score on a scale | 17.84 (17.62) | 17.84 (17.62)

17. Secondary Outcome: RSI Score by Subject
Description: Subject-reported outcome of RSI score.
  The Rhinosinusitis Symptom Inventory (RSI) scale ranges from 0 to 60. Higher scores indicate a worse outcome.
Time Frame: Day 180
Population: Number of units (sinus sides) analyzed represents number of participants with data evaluable.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 79 | 79
Number analyzed (sinus sides) | 77 | 77
score on a scale | 7.7 (7.84) | 7.7 (7.84)

18. Secondary Outcome: Implant Delivery Success by Clinical Investigators
Description: Number of subjects who underwent successful access and deployment of the PROPEL Contour Sinus Implant into the FSO. Delivery is considered successful if the procedure concludes with correct implant placement on the intended side, even if a second attempt to place the implant is necessary. An attempted deployment occurs when the investigator introduces the delivery system into the subject's nostril with the intent of placing an implant.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PROPEL Contour Sinus Implant
Number analyzed (Participants) | 80
Participants | 80

19. Post Hoc Outcome: Difference in FSO Patency at Day 45 - Baseline Zinreich's Modified Lund-Mackay Score ≥ 1 on Both Sides by Independent Reviewer Subgroup
Description: Side-to-side difference in FSO patency at Day 45 based on cross-sectional area of FSO by CT measurements performed by an independent, blinded reviewer, as assessed within the subgroup of participants with a baseline Zinreich's modified Lund-Mackay score ≥ 1 on both sides per independent, blinded reviewer.
Time Frame: Day 45
Population: Number of units (sinus sides) analyzed represents number of participants within the subgroup with data evaluable.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 46 | 46
Number analyzed (sinus sides) | 45 | 45
mm^2 | 14.98 (18.21) | 8.70 (12.88)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Test type: Superiority; p = 0.025, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Net) = 6.28, 95% CI 2-sided [0.8 to 11.7], Standard Deviation 18.12 — [estimate comment as in outcome 1, analysis 1]

20. Post Hoc Outcome: FSO Cross-sectional Area Change From Baseline on CT by an Independent, Blinded Reviewer - Baseline Zinreich's Modified Lund-Mackay Score ≥ 1 on Both Sides by Independent Reviewer Subgroup
Description: FSO cross-sectional area change from baseline to Day 45 and change from baseline to Day 180 per CT assessment performed by an independent, blinded reviewer, as assessed within the subgroup of participants with a baseline Zinreich's modified Lund-Mackay score ≥ 1 on both sides per independent, blinded reviewer. Cross-sectional area of FSO was measured via computer-assisted segmentation of CT images.
Time Frame: Baseline, Day 45, and Day 180
Population: Number of units (sinus sides) analyzed represents number of participants within the subgroup with data evaluable for the corresponding timepoint.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 46 | 46
Number analyzed (sinus sides) | 44 | 44
mm^2
  Change from baseline to Day 45 | 4.87 (9.59) | 0.89 (10.87)
  Change from baseline to Day 180: number analyzed (sinus sides) | 43 | 43
  Change from baseline to Day 180 | 4.29 (12.46) | 7.74 (16.12)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.04, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 3.98, 95% CI 2-sided [0.2 to 7.8], Standard Deviation 12.49 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.09, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Median Difference (Final Values) = -3.45, 95% CI 2-sided [-7.5 to 0.6], Standard Deviation 13.02 — [estimate comment as in outcome 2, analysis 2]

21. Post Hoc Outcome: CT Frontal Sinus Outflow Tract (FSOT) Volume by Blinded Reviewer - Baseline Zinreich's Modified Lund-Mackay Score ≥ 1 on Both Sides by Independent Reviewer Subgroup
Description: FSOT, referring to the region of the frontal sinus surrounding the FSO, bordered superiorly by the frontal infundibulum and inferiorly by the frontal recess, as assessed within the subgroup of participants with a baseline Zinreich's modified Lund-Mackay score ≥ 1 on both sides per independent, blinded reviewer. FSOT volume was measured via computer-assisted segmentation of CT images.
Time Frame: Days 45 and 180
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 46 | 46
Number analyzed (sinus sides) | 45 | 45
mm^3
  Day 45 | 306.06 (389.90) | 244.52 (394.58)
  Day 180: number analyzed (sinus sides) | 44 | 44
  Day 180 | 282.89 (394.99) | 334.86 (451.20)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.375, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 61.54, 95% CI 2-sided [-76.7 to 199.8], Standard Deviation 460.18 — Difference = PROPEL Contour Sinus Implant mean FSOT volume minus balloon sinus dilation alone mean FSOT volume
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.432, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -51.98, 95% CI 2-sided [-184.1 to 80.2], Standard Deviation 434.64 — Difference = PROPEL Contour Sinus Implant mean FSOT volume minus balloon sinus dilation alone mean FSOT volume

22. Post Hoc Outcome: CT FSO Minimum Diameter by Blinded Reviewer - Baseline Zinreich's Modified Lund-Mackay Score ≥ 1 on Both Sides by Independent Reviewer Subgroup
Description: CT FSO minimum diameter as assessed within the subgroup of participants with a baseline Zinreich's modified Lund-Mackay score ≥ 1 on both sides per independent, blinded reviewer. FSO minimum diameter was measured via computer-assisted segmentation of CT images.
Time Frame: Days 45 and 180
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: sinus sides
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
Number analyzed (Participants) | 46 | 46
Number analyzed (sinus sides) | 45 | 45
mm
  Day 45 | 2.31 (2.04) | 1.57 (1.60)
  Day 180: number analyzed (sinus sides) | 43 | 43
  Day 180 | 2.18 (2.07) | 2.33 (2.23)
Statistical Analysis 1: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 45; Test type: Superiority; p = 0.023, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [0.1 to 1.4], Standard Deviation 2.13 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: PROPEL Contour Sinus Implant vs Balloon Sinus Dilation Alone; Day 180; Test type: Superiority; p = 0.646, t-test, 2 sided — Paired; the threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.8 to 0.5], Standard Deviation 2.24 — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: From enrollment through Day 180 (end of study)
Description: A standard questionnaire was used to determine whether or not adverse events (AE) had occurred at the current follow-up visit or since the previous follow-up visit. Clinical investigators evaluated the occurrence of AEs excluding usual post-operative recovery signs and symptoms experienced by participants, unless corroborated by objective findings and/or requiring specific medical or therapeutic interventions.
Groups:
- PROPEL Contour Sinus Implant: All sinuses exposed to the PROPEL Contour Sinus Implant
- Balloon Sinus Dilation Alone: All sinuses that were not exposed to the PROPEL Contour Sinus Implant.
Arm/Group | PROPEL Contour Sinus Implant | Balloon Sinus Dilation Alone
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/80 | 1/80
Other Adverse Events (participants affected / at risk) | 15/80 | 16/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PROPEL Contour Sinus Implant (N=80) | Balloon Sinus Dilation Alone (N=80)
Loss of balance (Nervous system disorders) | 1 | 1 — Participant reported losing his balance while moving machinery down a ramp, resulting in a fall and bruising to his ribs, knee, and lower back. Loss of balance cannot be localized to a side, so each instance is represented in both arms.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PROPEL Contour Sinus Implant (N=80) | Balloon Sinus Dilation Alone (N=80)
Chronic sinusitis (Infections and infestations) | 11 | 13 — Number affected reflects number of participants with at least once instance of the adverse event localized to either the treatment or control side.
COVID-19 (Infections and infestations) | 12 | 12 — Number affected reflects number of participants with at least once instance of the adverse event. COVID-19 cannot be localized to a side, so each instance is represented in both arms.

LIMITATIONS AND CAVEATS:
Per study eligibility criteria, participants were required to have a Lund-Mackay score ≥1 on both frontal sinus sides at baseline as assessed by clinical investigators. Only roughly half of participants met this criteria per independent, blinded review. This may confound results, as a Lund-Mackay score of ≥1 indicates CT evidence of sinonasal inflammation and is recommended as a precondition for surgery in the International Consensus Statement on Allergy and Rhinology: Rhinosinusitis 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT04858802/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT04858802/SAP_001.pdf